## Cannabis Edibles Packaging Imagery Experiment

IRB Approved Date 02APR2024

NCT06358144

## Adult Consent Form Cannabis Edibles Packaging Imagery Experiment IRB00111438

## Perceptions of Marijuana Edibles and their Packaging (Version 2)

You are invited to complete a survey as part of a research study being conducted by Wake Forest University School of Medicine. The goal of the survey is to understand what adults think about marijuana edible products and their packaging. Marijuana edibles are food products that contain marijuana. You will answer a few questions to determine if you qualify for the study. You do not need to be a user of marijuana to take part in this study. If you qualify for the study, in the survey you will be shown four packages of marijuana edibles and asked to answer questions to give your opinion on each one. We will also ask you some information about yourself. The survey will take about 15 minutes to complete. We expect that about 1,250 people will take this survey.

There is no cost to you to take the survey. Upon completion of the survey, you will be provided with compensation as agreed upon with your panel. Your participation is completely voluntary. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. You may choose not to take part in the study or leave the study at any time.

You are not expected to receive any direct benefit from taking part in this research study. We hope that the information learned from this study will benefit other people in the future. The study is not intended to provide treatment for any disease or condition. The alternative to participating in the study is to not participate.

The risk of harm or discomfort that may happen as a result of taking part in this research is not expected to be more than in daily life or from routine physical or psychological examinations or tests. There is a slight risk of breach of confidentiality. We will do our best to protect your confidential information by not collecting any information that could identify you and by keeping records secure, allowing only authorized persons to have access. No reference to any individual will appear in reports, presentations, or publications that may arise from the study.

| The person in charge of this study is Beth Reboussin, PhD. If you have any questions, suggestions, or |
|---|
| concerns regarding this study, or if you wish to withdraw from the study, please contact Dr. Reboussin at |
| . If you have any questions, suggestions, or concerns about your rights as a |
| volunteer in this research, please contact the Wake Forest Institutional Review Board at |
| Wake Forest Research Subject Advocate at . |

A Certificate of Confidentiality from the National Institutes of Health covers this research. This means that the researchers cannot release any information that may identify you in any legal action unless it is required by law or you grant permission. This protection applies to federal, state, or local civil, criminal, administrative, legislative, or other proceedings. There are two exceptions: First, we must follow laws that require the reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. Second, you can willingly release information about your involvement in this research. To find out more about Certificates of Confidentiality, visit: <a href="https://grants.nih.gov/policy/humansubjects/coc.htm">https://grants.nih.gov/policy/humansubjects/coc.htm</a>.

Checking the box below indicates that:

- You have read the above information
- You voluntarily agree to participate
- You are at least 18 years of age

| Please check "I agree" if you would like to participate |
|---------------------------------------------------------|
| ☐ I agree |
| ☐ I do not agree |
| - |

Version: 1 (3/7/2024)